CLINICAL TRIAL: NCT03168919
Title: Image-Based Quantitative Assessment of Acute Radiation-Induced Changes in Glioma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI is leaving institution
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Asim Bag, Associate Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: F160324004
Record Dates: First submitted 2017-04-28; First posted 2017-05-30 (Actual); Results first posted 2019-07-02 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — Temozolomide

STUDY DESIGN:
Intervention Model Description: One arm study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Chemoradiation with MRI assessment (Experimental): This study has only one arm. The eligible subjects will receive standard of care fractionated radiation therapy along with concomitant temozolomide, which will NOT be changed based on the MRI scans obtained as a part of this study. There is no control or sham group.
  Interventions: Radiation: Fractionated Radiation; Drug: Temozolomide; Device: MRI

INTERVENTIONS:
Radiation: Fractionated Radiation — Standard of care fractionated radiation therapy will be given to the tumor.
Drug: Temozolomide — Standard of care temozolomide will be given along with radiation therapy
  Other Names: Temodar
Device: MRI — Four MRI scan will be performed according to the protocol. The first one will be obtained before start of radiation therapy, the second MRI will be obtained after completion of 20 +/- 4 Gy, the third MRI will be obtained after completion of 40 +/- 4 Gy, and the final MRI will be obtained after completion of the radiation therapy.
  Other Names: Multi parametric MRI including MR spectroscopy

SUMMARY:
The overall goal of this study is to determine if quantitative imaging techniques can be used to detect dynamic changes of morphology and different physiologic properties of the tumor during and after completion of radiation treatment and to predict site and time of radiation.

DETAILED DESCRIPTION:
Once eligibility criteria have been assessed and the informed consent is obtained, participants will undergo a screening process to further ensure eligibility. Screening prior to registration will comprise a review of pathology reports, postoperative magnetic resonance Imaging (MRI) images, operative reports, and medical history; general physical and neurologic exams; routine blood work; and urine pregnancy test for women of childbearing age.

The study is intended to evaluate the response of radiation treatment (RT). The consent process will be performed between the surgery and the start of RT. RT will be prescribed as per the discretion of the treating radiation oncologist as per the University of Alabama at Birmingham Department of Radiation Oncology treatment protocol in combination with temozolomide.

MRIs will be obtained before start of RT, after completion of 20 +/- 4 Gy. after completion of 40+/- 4 Gy and after the entire radiation treatment. Conventional MRIs including perfusion sequences and whole brain spectroscopy will be performed as a part of the research study. The data obtained from this research studies will not be used for clinical management.

Volumes of the enhancing component, non enhancing component, choline/N-acetyl aspartate (Cho/NAA) will be measure before, during and after RT as described before. Cerebral blood volume (CBV) of the tumor will also be calculated from perfusion imaging at each time point. Apparent diffusion co-efficient (ADC) of the tumor will be calculated from the diffusion imaging.

All the patients will be followed up with imaging and will be treated as per the standard of care. Patients will return for clinical evaluation and standard of care imaging approximately 4 weeks from the completion of the radiation therapy. After that, all the patients will be treated with standard of care maintenance temozolomide therapy and will return every 2-3 months for clinical evaluation and standard of care imaging.

At the time of recurrence, the recurrence site will be assessed and will be compared with the imaging parameters obtained during radiation treatment. Time to recurrence will also be calculated and will be correlated with the imaging parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed glioma, based on pathology confirmation;
2. At least 8 cm3 of residual enhancing tumor after surgery or significant visible tumor (As seen on immediate postoperative scan);
3. Scheduled to receive standard fractionated RT with concomitant temozolomide therapy;
4. Karnofsky Performance Score > 60.

Exclusion Criteria:

1. Scheduled to receive investigational chemotherapy, immunotherapy, or any other investigational agents;
2. Placement of GLIADEL® wafer in the resection cavity;
3. Significant amount of hemorrhage within the resection cavity (seen on immediate post-operative scan);
4. A large peritumoral infraction related to surgery (identified by new confluent diffusion restriction);
5. Not suitable to undergo MRI or use the MRI contrast agent (GFR<30 mL/min/1.73 m2); or the patient has known anaphylactic reaction to gadolinium based contrast agents.
6. Presence of serious systemic illness, including: uncontrolled infection, uncontrolled malignancy, significant renal disease, or psychiatric/social situations, which might impact the survival endpoint of the study or limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asim Bag, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 10/2016 through 3/2018
  Location: The subjects were identified from the hospital during the admission for resection of the tumor. They were recruited from the clinic of the radiation oncologists and/or neurosurgeons.
Pre-assignment Details: Subject #2: Voluntary withdrawal. Subject #5: Voluntary withdrawal.
Period: Overall Study
Arm/Group | Chemoradiation With MRI Assessment
Started | 5
Completed | 3
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Five subjects participated in the baseline. Two of them voluntarily withdrew. Only 3 subjects completed the treatment.
Arm/Group | Chemoradiation With MRI Assessment
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 62.8 [53 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
Glioblastoma Diagnosis [Count of Participants; unit: Participants] | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Changes of the Chemical Environment of the Tumor
Description: Multiple MRI techniques will be used to assess chemical environment (Cho/NAA) of the tumor during the course of fractionated radiation treatment.
Time Frame: From Baseline to 6 weeks.
Population: The number of participants dropped from 5 to 3 because 2 participants withdrew from the study. The chemical evaluation could not be evaluated due to poor quality imaging.
Arm/Group | Chemoradiation With MRI Assessment
Number analyzed (Participants) | 0
Statistical Analysis 1: Comparison: Chemoradiation With MRI Assessment; The baseline and the end of therapy MRI parameters are compared; Test type: Other — Comparison; Due to very small accrual, the statistical analysis couln't be performed

2. Secondary Outcome: Changes of Tumor Cellularity
Description: Diffusion MRI will be used for assessment of measures tumor cellularity (with minimum apparent diffusion co-efficent, ADC) during the course of fractionated radiation treatment.
Time Frame: From baseline to 6 weeks
Population: Only 3 subjects completed the treatment.
Measure: Mean (Full Range); unit: mm^2/sec
Groups:
- Chemoradiation Arm: Diffuion MRI was performed before, during and after completion of radiation
Arm/Group | Chemoradiation Arm
Number analyzed (Participants) | 3
mm^2/sec
  Baseline | 0.000675 [0.000580 to 0.000821]
  Early in therapy (At 2 weeks in therapy) | 0.000798 [0.000642 to 0.000984]
  Late therapy (At 4 weeks in therapy) | 0.000842 [0.000675 to 0.0013]
  At completion (At 6 weeks from baseline) | 0.001144 [0.000753 to 0.0018]

3. Secondary Outcome: Changes of Tumor Volume
Description: MRI will be used for assessment of measures tumor volume.
Time Frame: From baseline Up to 6 weeks
Population: Measurements performed only in 2 subjects .
Measure: Mean (Full Range); unit: cm3
Groups:
- Chemoradiation Arm: Volumetric MRI was performed before, during and after completion of radiation
Arm/Group | Chemoradiation Arm
Number analyzed (Participants) | 2
cm3
  Baseline | 6.1 [4.6 to 8]
  Early in therapy (At 2 weeks in therapy) | 3.79 [1.5 to 6.5]
  Late therapy (At 4 weeks in therapy) | 2.66 [0.49 to 4.6]
  At completion (At 6 weeks from baseline) | 2.16 [0.52 to 3.8]

4. Secondary Outcome: Changes of Tumor Angiogenesis
Description: Perfusion MRI will be used for assessment of tumor angiogenesis (with median normalized cerbral blood volume, nCBV) during the course of fractionated radiation treatment.
Time Frame: From baseline to 6 weeks
Population: Results of only 2 subjects was included.
Measure: Mean (Full Range); unit: mL/100 gm of brain tissue
Groups:
- Chemoradiation Arm: Perfusion MRI was performed before, during and after completion of radiation
Arm/Group | Chemoradiation Arm
Number analyzed (Participants) | 2
mL/100 gm of brain tissue
  baseline | 3.78 [0.9 to 5.34]
  Early in therapy (At 2 weeks in therapy) | 3.35 [1.3 to 5.4]
  Late therapy (At 4 weeks in therapy) | 1.58 [1.05 to 2.3]
  At completion (At 6 weeks from baseline) | 1.2 [0.21 to 2.2]

5. Other Pre Specified Outcome: Time to Progression
Description: Percentage change of the Cho/NAA, ADC and nCBV from baseline to the end of radiation therapy, RT will be used for assessment of time to progression.
Time Frame: From Baseline through 24 months.
Measure: Mean (Full Range); unit: days
Groups:
- Chemoradiation Arm: Only 3 subjects were imaged
Arm/Group | Chemoradiation Arm
Number analyzed (Participants) | 3
days | 465 [252 to 820]

ADVERSE EVENTS:
Time Frame: 1 year 6 months
Arm/Group | Chemoradiation With MRI Assessment
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
The study enrollment was much less than anticipated. With only 5 subjects in the study, it is difficult to make a meaningful conclusion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-14): https://cdn.clinicaltrials.gov/large-docs/19/NCT03168919/Prot_SAP_000.pdf